CLINICAL TRIAL: NCT04786717
Title: Restoration of Lumbopelvic Movement Control: Effect of Injury History, and the Role of Cortical Control and Its Practical Application(1)
Brief Title: Lumbopelvic Movement Control: Effect of Injury History, and the Role of Cortical Control and Its Practical Application 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yi-Fen Shih, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YM110027E(1)
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Biomechanical Phenomena
Keywords: back pain history; deep squat; movement control; cortical control; imagery training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- core muscle training (Experimental): Training the endurance of the core muscle.
  Interventions: Other: core muscle training
- movement control training (Experimental): Based from the initial test, the subjects will receive lumbar movement control exercise. They will perform each lumbar movement control exercise in different position.
  Interventions: Other: movement control training
- combined imagery and movement control training (Experimental): The intervention of this group is mostly same as the movement control training group. The different part is that the first 3 times of the movement will be practiced through image training, and the subjects will practice the real movement in the rest of 7 times.
  Interventions: Other: combined imagery and movement control training

INTERVENTIONS:
Other: core muscle training — The intervention of this group will focus on training the endurance of the core muscle.
  Arms: core muscle training
Other: movement control training — Based from the initial test, the subjects will receive either lumbar flexion control exercise or lumbar extension control exercise. They will perform each lumbar movement control exercise in different position. Starting from the lying position, then progressing to sitting, standing with support, and the last level will be standing without support. Each set of movement will be practiced 10 times, totally 10 sets. It will take approximately 5~8 minutes to finish each movement. The subjects will learn 5~8 types of the movement every week.
  Arms: movement control training
Other: combined imagery and movement control training — The intervention of this group is mostly same as the movement control training group. The different part is that the first 3 times of the movement will be practiced through image training, so the subjects will not have any real movement, and the last 7 times they will perform the lumbar motor control exercise literally. Each set of movement will be practiced 10 times, totally 10 sets. It will take approximately 5~8 minutes to finish each movement. The subjects will learn 5~8 types of the movement every week.
  Arms: combined imagery and movement control training

SUMMARY:
Lumbopelvic movement control is crucial for movement stability during weight loading training, and also an important risk factor for the occurrence and recurrence of low back pain (LBP). Previous studies indicated that athletes with LBP had poorer lumbopelvic movement control, and the deficits in lumbopelvic control could be remained after LBP remission. However, there has been no study investigating the effect of LBP history (LBPH) on the performance of the loaded squatting task, and lumbopelvic movement control in people who practice regular weight training.

Therefore, the aims of this study are to examine the differences in lumbopelvic movement control, kinematics and muscle activation during the loaded squatting task in weight training practitioners with LBP, LBPH, and asymptomatic controls, to compare the cortical control mechanisms between 3 types of motor control training strategies, and to investigate the intervention effect of motor control training on restoring the lumbopelvic movement control and squatting performance.

DETAILED DESCRIPTION:
Lumbopelvic movement control is crucial for movement stability during high weight loading training, and also an important risk factor for the occurrence and recurrence of low back pain (LBP). Previous studies indicated that athletes with LBP had poorer lumbopelvic movement control, and for those athletes who have recovered from LBP, some research data still showed that poor lumbopelvic control remained. However, there has been no study investigating the effect of LBP history (LBPH) on the performance of the loaded squatting task, and lumbopelvic movement control in people who practice regular weight training.

Therefore, the aims of this study are to examine the differences in lumbopelvic movement control, kinematics and muscle activation during the loaded squatting task in weight training practitioners with LBP, LBPH, and asymptomatic controls. In the next part of the study, investigators will further investigate the intervention effect of motor control training on restoring the lumbopelvic movement control and squatting performance. Methods: This is an exploratory, cross-sectional, and intervention study. First part: investigators plan to recruit 15 participants between 20-40 years old, practicing loaded squatting for 1 day a week for at least one year, and having LBPH; 15 matched participants with current LBP, and 15 controls for the study. All subjects will undergo a series of squatting task (4 X 10 repetitions) and the kinematics and muscle activation of the rectus abdominus, transverse abdominus/internal obliqus, eractor spinae, and gluteus maximus will be recorded and analyzed using Noraxon myoRESEARCH (Noraxon U.S.A., Inc., Scottsdale, AZ, USA). A set of lumbopelvic movement control tests will also be conducted. The kinematics, muscle activation, and movement control test scores will be compared between groups. The second part, investigators plan to recruit 45 weight training practitioners with LBPH, randomized into three groups (core muscle training, movement control training, combined imagery and movement control training), and compare the effect of 4-week training on squatting performance and lumbopelvic movement control. Statistical analysis: Comparisons of all continuous variables are performed using the analysis of variance (ANOVA), and the intervention effect will be assessed using the repeated measures ANOVA. Chi squared test is used to examine the group differences in lumbopelvic movement control testing. The significance level is set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

Frequency of weight loading squatting training:

1. At least 1 time/week, at least 1 year.

LBP group:

1. Present symptoms from T12 to the upper buttock
2. Numerical rating scale (NRS) score ≥ 3/10
3. Present episode of LBP lasting > 24 hours

LBPH group:

1. Previous symptoms from T12 to the upper buttock
2. Presently in symptom remission
3. At least 2 episodes of LBP in the past 1 year, each lasting > 24 hours, and following a period of at least 2~4 weeks pain-free, OR at least 1 episode of LBP, each lasting 2 months.

Asymptomatic controls:

1. Without any history of LBP that limited their function or required treatment from a health professional in the past 2 years.

Exclusion Criteria:

1. Inability to perform parallel-squat due to LBP
2. Pain and ROM limitation in lower extremities
3. LBP due to traumatic injury
4. Previous spine surgery
5. Spinal deformities: HIVD, spondylosis, scoliosis, spinal stenosis
6. Neurological sign, and radiating pain to lower extremities
7. Systematic disease: rheumatoid arthritis

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2021-11-14 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Lumbopelvic kinematics | pre-intervention
  The investigator will place three markers at subjects' 1st lumbar vertebrae, 2nd sacrum vertebrae, and lateral side of left greater trochanter. The investigator will record the track of each marker through the video system(Noraxon myoVIDEOTM, Noraxon USA Inc., USA) while the subject is squatting. According to the record, the investigator will analyze the angles between 1st lumbar vertebrae and 2nd sacrum vertebrae which are the lumbar flexion angles and the lumbar extension angles.
Lumbopelvic kinematics | after 4 weeks of intervention
  The investigator will place three markers at subjects' 1st lumbar vertebrae, 2nd sacrum vertebrae, and lateral side of left greater trochanter. The investigator will record the track of each marker through the video system(Noraxon myoVIDEOTM, Noraxon USA Inc., USA) while the subject is squatting. According to the record, the investigator will analyze the angles between 1st lumbar vertebrae and 2nd sacrum vertebrae which are the lumbar flexion angles and the lumbar extension angles.
Hip kinematics | pre-intervention
  The investigator will place three markers at subjects' 1st lumbar vertebrae, 2nd sacrum vertebrae, and lateral side of left greater trochanter. The investigator will record the track of each marker through the video system(Noraxon myoVIDEOTM, Noraxon USA Inc., USA) while the subject is squatting. According to the record, the investigator will analyze the angles between 2nd sacrum vertebrae and greater trochanter which are the hip flexion angles and the hip extension angles.
Hip kinematics | after 4 weeks of intervention
  The investigator will place three markers at subjects' 1st lumbar vertebrae, 2nd sacrum vertebrae, and lateral side of left greater trochanter. The investigator will record the track of each marker through the video system(Noraxon myoVIDEOTM, Noraxon USA Inc., USA) while the subject is squatting. According to the record, the investigator will analyze the angles between 2nd sacrum vertebrae and greater trochanter which are the hip flexion angles and the hip extension angles.
Muscle activation | pre-intervention
  The investigator will record the muscle activation of erector spinae, rectus abdominus, internal obliques, and gluteus maximus through the electromyography (Noraxon TeleMyo sEMG System, Noraxon USA Inc., USA)
Muscle activation | after 4 weeks of intervention
  The investigator will record the muscle activation of erector spinae, rectus abdominus, internal obliques, and gluteus maximus through the electromyography (Noraxon TeleMyo sEMG System, Noraxon USA Inc., USA)
Lumbopelvic control ability | pre-intervention
  Using lumbar motor control test battery to test the stability of subjects' lumbar. This test battery is consisted of 10 motor control test based from previous studies. If the subjects complete the test successfully, they will get 1 point in each test, otherwise they may not get any points. Therefore, the minimum of the scale is 0 point, and the maximum is 10 points, and the higher scores mean the subjects can control their lumbar vertebrae much better.
Lumbopelvic control ability | after 4 weeks of intervention
  Using lumbar motor control test battery to test the stability of subjects' lumbar. This test battery is consisted of 10 motor control test based from previous studies. If the subjects complete the test successfully, they will get 1 point in each test, otherwise they may not get any points. Therefore, the minimum of the scale is 0 point, and the maximum is 10 points, and the higher scores mean the subjects can control their lumbar vertebrae much better.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Fen Shih, PhD, Study Director — Department of Physical Therapy and Assistive Technology, National Yang-Ming Chiao-Tung University
Locations (1):
- National Yang Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No